CLINICAL TRIAL: NCT03783026
Title: A Phase 4, Multicenter, Single-Arm, Open-Label Study to Evaluate the Impact of Apremilast (CC-10004) on MRI Outcomes in Subjects With Active Psoriatic Arthritis
Brief Title: A Study to Evaluate the Impact of Apremilast on Magnetic Resonance Imaging (MRI) Outcomes in Adults With Psoriatic Arthritis
Acronym: MOSAIC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-10004-PSA-014; U1111-1223-9823 (Registry Identifier: WHO); 2018-002748-10 (EudraCT Number)
Record Dates: First submitted 2018-12-14; First posted 2018-12-20 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; CC-10004; MRI; apremilast
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — apremilast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Apremilast (Experimental): Participants will receive apremilast 30 mg twice a day for 48 weeks.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Tablets for oral administration
  Other Names: CC-10004; Otezla®

SUMMARY:
This study is designed to assess the efficacy of apremilast, either in monotherapy or with stable methotrexate, on imaging outcomes in adults with active psoriatic arthritis with less than 5 years of disease duration (since diagnosis), and who are naïve to biologic therapies.

DETAILED DESCRIPTION:
This study consists of 3 phases:

* Screening Phase - up to 4 weeks
* Single-arm, Open-label Treatment Phase - Weeks 0 to 48

  * Participants will receive apremilast 30 mg BID (after a 5-day titration period) for the entire duration of this phase.
  * MRI of the most affected hand and whole body MRI (WB-MRI) will be performed at weeks 0, 24, and 48.
  * The hand with the greater inflammatory burden of swollen joints and/or dactylitis will be considered as the most affected hand. If both hands are equally affected, the dominant hand will be designated as the index hand.
* Observational Follow-up Phase - 4 Weeks

  * All participants who complete the study or discontinue early will participate in the 4-week Post-Treatment Observational Follow-up Phase.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Males or females, aged ≥ 18 years at time of consent
2. For all regions, the local Regulatory Label for treatment with apremilast must be followed.
3. Must understand and voluntarily sign an informed consent document prior to any study related assessments/procedures being conducted
4. Able to adhere to the study visit schedule and other protocol requirements
5. Have a documented diagnosis of PsA of ≥ 3 months AND ≤ 5 years in duration, meeting the Classification Criteria for Psoriatic Arthritis (CASPAR) at the time of Screening Visit
6. Have ≥ 3 swollen AND ≥ 3 tender joints, with hand involvement (defined as ≥ 1 swollen joint or dactylitis [each clinically active joint of a dactylitic digit is counted as one joint]).
7. Have at least 1 active enthesitis site (one of the Spondyloarthritis Research Consortium of Canada [SPARCC] or Leeds Enthesitis Index [LEI] sites)
8. Must not have been treated previously with a tumor necrosis factor (TNF) blocker or other biologic drug for PsA treatment
9. Must not have been treated with more than 2 conventional synthetic disease-modifying antirheumatic drugs (csDMARDs)
10. Subjects taking csDMARDs, with the exception of methotrexate (MTX), cyclosporine, or leflunomide (LEF), do not require a washout period. However, they must discontinue the csDMARD treatment at least one day prior to their Baseline Visit (ie, Visit 2, Day 1)
11. Subjects who have been previously treated with MTX for < 6 months and who are not on stable doses for at least 3 months will require a 28-day washout prior to the Baseline Visit to participate in the study
12. Subjects who have been previously treated with LEF will require a 12-week washout prior to the Baseline Visit, or treatment with cholestyramine, per LEF prescribing label (ie, 8 g cholestyramine 3 times daily for 11 days)
13. Subjects who have been previously treated with cyclosporine will require a 28-day washout prior to the Baseline Visit to participate in the study
14. If taking MTX (≤ 25 mg/week), continuity of treatment will be allowed if duration of treatment is ≥ 6 months and on a stable dose for at least 3 months prior to the Baseline Visit
15. If taking oral glucocorticoids, must be on a stable dose of prednisone ≤ 10 mg/day or equivalent for at least 4 weeks prior to the Baseline Visit
16. If taking nonsteroidal anti-inflammatory drugs (NSAIDs) or narcotic analgesics, must be on stable dose for at least 4 weeks prior to Baseline Visit
17. A female of childbearing potential (FCBP) must have a negative pregnancy test at screening and baseline. While on investigational product (IP) and for at least 28 days after taking the last dose of IP, a FCBP who engages in activity in which conception is possible must use one of the approved contraceptive options described below:

    Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device; tubal ligation; or partner's vasectomy; OR Option 2: Male or female condom (latex condom or non-latex condom NOT made out of natural [animal] membrane [for example, polyurethane]); PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.
18. Must be in general good health (except for PsA) as judged by the investigator, based on medical history, physical examination, and clinical laboratories. (Note: The definition of good health means a subject does not have uncontrolled significant comorbid conditions).

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Contraindication to MRI examination including, but not limited to, intracranial metal clips, heart pacemakers, insulin pumps, implanted hearing aids, neurostimulators, metal hip replacements, profound claustrophobia or inability to lie in the MRI machine in an appropriate position to obtain quality images, history of hypersensitivity to gadolinium contrast agent
2. Severe renal impairment (creatinine clearance of less than 30 mL per minute estimated by the Cockroft-Gault equation), which would prevent the use of gadolinium enhancement
3. History of clinically significant (as determined by the investigator) cardiac, endocrine, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major uncontrolled disease
4. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
5. Prior history of suicide attempt at any time in the subject's lifetime prior to signing the informed consent, or major psychiatric illness requiring hospitalization within the last 3 years prior to signing the informed consent.
6. Pregnant or breast feeding
7. Active substance abuse or a history of substance abuse within 6 months prior to screening
8. History of allergy or hypersensitivity to any component of the IP
9. History of rare hereditary problems of galactose intolerance, lapp lactase deficiency or glucose-galactose malabsorption
10. History of positive human immunodeficiency virus (HIV), or congenital or acquired immunodeficiency (eg, Common Variable Immunodeficiency Disease)
11. Active tuberculosis or a history of incompletely treated tuberculosis
12. Bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of screening. Any treatment for such infections must have been completed and the infection cured, at least 4 weeks prior to screening and no new or recurrent infections prior to the Baseline Visit
13. Malignancy or history of malignancy or myeloproliferative or lymphoproliferative disease within the past 3 years, except for treated (ie, cured) basal cell or squamous cell in situ skin carcinomas;
14. Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following Baseline Visit
15. Rheumatic autoimmune disease other than PsA, including, but not limited to: systemic lupus erythematosus, mixed connective tissue disease, scleroderma, polymyositis, or fibromyalgia
16. Prior history of or current inflammatory joint disease other than PsA (eg, gout, reactive arthritis, rheumatoid arthritis, ankylosing spondylitis, Lyme disease), which confounds the ability to interpret data from the study
17. Prior treatment with any biologic DMARD
18. Prior treatment with more than 2 csDMARDs
19. Use of the following systemic therapy(ies) within 28 days of the Baseline Visit: cyclosporine or other calcineurin inhibitors, glucocorticoids exceeding 10 mg daily prednisone equivalent, as well as mycophenolate.
20. Use of MTX within 4 weeks of the Baseline Visit, unless subject is on stable doses for at least 3 months and total treatment duration with MTX is ≥ 6 months
21. Use of LEF within 12 weeks of the Baseline Visit, unless subject has taken cholestyramine, 8 g three times daily 11 days after stopping LEF
22. Previous treatment with a Janus kinase (JAK) inhibitor (including tyrosine kinase 2 [TYK2] inhibitor)
23. Prior treatment with apremilast, or participation in a clinical study involving apremilast
24. Use of intra-articular (IA) glucocorticoid injection within 8 weeks before the Baseline Visit.
25. Use of any investigational drug within 4 weeks of the Baseline Visit, or 5 pharmacokinetic/pharmacodynamic half-lives, if known (whichever is longer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (36):
- United States (7):
  - The Doctors of Saint John's Medical Group, Santa Monica, California
  - Inland Rheumatology Clinical Trials Inc, Upland, California
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - Integral Rheumatology and Immunology Specialists, Plantation, Florida
  - NYU Langone Medical Center, New York, New York
  - Austin Regional Clinic, Austin, Texas
  - Swedish Medical Center, Seattle, Washington
- Medizinische Universitat Wien, Vienna, Austria
- UZ Leuven, Leuven, Belgium
- Canada (4):
  - University of Calgary - Cumming School of Medicine, Calgary, Alberta
  - Alberta Rheumatology, Edmonton, Alberta
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - G.R.M.O. (Groupe de recherche en maladies osseuses) Inc., Québec, Quebec
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - Frederiksberg Hospital, Frederiksberg
  - Copenhagen University Hospital Rigshospitalet, Glostrup Municipality
- Germany (4):
  - Universitaetsklinikum Bonn, Bonn
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Johann Wolfgang Goethe University Hospital, Frankfurt am Main
  - Universitaetsklinikum Tuebingen, Tübingen
- Italy (2):
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele Ospedale Vittorio Emanuele, Catania
  - Azienda Ospedaliera Regionale San Carlo, Potenza/Matera
- Russia (5):
  - Udmurt Republic Republican Clinical Diagnostic Center, Izhevsk
  - Research Institute of Rheumatology named after V.A.Nasonova, Moscow
  - LLC Medical Center Zdorovaya Semiya, Novosibirsk
  - Mechnikov North-Western State Medical University, Saint Petersburg
  - Regional Clinical Hospital No 1 - Tyumen, Tyumen
- Spain (3):
  - Hospital Virgen de Macarena, Seville, Andalusia
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital La Paz, Madrid
- Switzerland (3):
  - Kantonsspital Aarau - KSA, Aarau
  - Hopital Universitaire Genevois - Beau-Sejour Hospital, Geneva
  - Kantonsspital St Gallen, Sankt Gallen
- United Kingdom (3):
  - NHS Lothian, Western General Hospital, Edinburgh
  - The Leeds Teaching Hospitals NHS Trust - Chapel Allerton Hospital, Leeds
  - Southampton University Hospitals NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Background] Ostergaard M, Boesen M, Maksymowych WP, Lambert RG, Bubb MR, Kubassova O, Valenzuela G, Reddy J, Colgan S, Klyachkin Y, Deignan C, Zhou Z, Amouzadeh H, Mease PJ. Effect of apremilast on hand and whole-body MRI assessments of inflammation in patients with psoriatic arthritis (MOSAIC): a phase 4, multicentre, single-arm, open-label study. Lancet Rheumatol. 2025 Feb;7(2):e118-e126. doi: 10.1016/S2665-9913(24)00232-7. Epub 2024 Oct 30. PMID 39488216
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 43 centers in Austria, Belgium, Canada, Denmark, Germany, Italy, Russia, Spain, Switzerland, United Kingdom, and the United States.
Pre-assignment Details: This was a single-arm, open-label study to evaluate the impact of apremilast on magnetic resonance imaging (MRI) outcomes in adults with psoriatic arthritis (PsA). The study consisted of a 48-week treatment phase, and an observational 4-week follow-up phase.
Groups:
- Apremilast: Participants received apremilast 30 mg twice a day for 48 weeks.
Period: Treatment Phase
Arm/Group | Apremilast
Started | 123
Received Apremilast | 122
Completed (Completed Treatment Phase) | 80
Not Completed | 43
Not completed — Adverse Event | 15
Not completed — Lack of Efficacy | 11
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 2
Not completed — Protocol Deviation | 8
Not completed — Did Not Receive Treatment | 1
Period: Observational Follow-up Phase
Arm/Group | Apremilast
Started (Per protocol, all participants who terminated early or completed the study treatment were asked to continue the 4-week post-treatment observational follow-up. Eleven participants did not enter the follow-up phase.) | 111
Completed | 108
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Apremilast
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (12.89)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 111
  ≥ 65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 111
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 117
  More than one race | 0
  Unknown or Not Reported | 2
Duration of Psoriatic Arthritis [Mean (Standard Deviation); unit: years] — From time of diagnosis to time the informed consent was signed. Population: The full analysis set includes all participants who were enrolled, and excludes participants who did not receive any study drug.
  years
    number analyzed (Participants) | 122
    (all) | 1.9 (1.66)
Synovitis Score Assessed by PsAMRIS [Mean (Standard Deviation); unit: score on a scale] — The Outcome Measures in Rheumatology (OMERACT) Psoriatic Arthritis Magnetic Resonance Imaging Score (PsAMRIS) scoring system assesses metacarpophalangeal (MCP), proximal interphalangeal (PIP), and distal interphalangeal (DIP) joints of fingers 2 to 5 of the most affected hand (the hand with the greater inflammatory burden of swollen joints and/or dactylitis).
  Synovitis was scored from 0 to 3 at MCP, PIP and DIP joints of fingers 2 to 5 (total of 12 joints), where score 0 is normal, and score 1-3 is mild, moderate, severe, respectively. The overall score ranges from 0 (normal) to 36 (severe). Population: Full analysis set participants with available data.
  score on a scale
    number analyzed (Participants) | 115
    (all) | 6.13 (5.121)
Tenosynovitis Score Assessed by PsAMRIS [Mean (Standard Deviation); unit: score on a scale] — Tenosynovitis is inflammation of the protective sheath (synovial membrane) that surrounds tendons.
  The OMERACT PsAMRIS scoring system assesses metacarpophalangeal (MCP), proximal interphalangeal (PIP), and distal interphalangeal (DIP) joints of fingers 2 to 5 of the most affected hand (the hand with the greater inflammatory burden of swollen joints and/or dactylitis).
  Flexor tenosynovitis was scored from 0 to 3 at 12 joints, where 0: none; 1: < 1/2 tendon thickness; 2: ≥ 1/2 and < 1 tendon thickness; 3: ≥ 1 tendon thickness. The overall score ranges from 0 (none) to 36 (severe). Population: Full analysis set participants with available data.
  score on a scale
    number analyzed (Participants) | 115
    (all) | 1.70 (3.268)
Bone Marrow Edema Score Assessed by PsAMRIS [Mean (Standard Deviation); unit: score on a scale] — Bone marrow edema (BME) is a buildup of fluid inside the bones. The OMERACT PsAMRIS scoring system assesses BME at the proximal and distal regions of MCP, PIP, and DIP joints of fingers 2 to 5 of the most affected hand. BME was assessed on a scale of 0-3 based on the proportion of bone with edema, compared to the assessed bone volume (articular surface to a depth of 1 cm), judged on all available images; where 0: no edema; 1: 1-33% of bone edema; 2: 34-66% of bone edema; 3: 67-100% of bone edema. The overall score ranges from 0 (none) to 72 (severe). Population: Full analysis set participants with available data.
  score on a scale
    number analyzed (Participants) | 114
    (all) | 3.02 (4.942)
Composite Score of BME, Synovitis, and Tenosynovitis Assessed by PsAMRIS [Mean (Standard Deviation); unit: score on a scale] — The OMERACT PsAMRIS scoring system assesses MCP, PIP, and DIP joints of fingers 2 to 5 of the most affected hand.
  Synovitis, flexor tenosynovitis, and bone edema were each scored from 0 (none/normal) to 3 (severe) at each joint. The total scores for synovitis and tenosynovitis range from 0 to 36 and the total score for BME ranges from 0 to 72.
  The PsAMRIS composite inflammation score is calculated as:
  BME score + 2 × synovitis score + 2 × tenosynovitis score. The score ranges from 0 (normal) to 216 (severe). Population: Full analysis set participants with available data.
  score on a scale
    number analyzed (Participants) | 114
    (all) | 18.51 (17.849)
Composite Score of BME and Synovitis Assessed by PsAMRIS [Mean (Standard Deviation); unit: score on a scale] — The OMERACT PsAMRIS scoring system assesses MCP, PIP, and DIP joints of fingers 2 to 5 of the most affected hand.
  Synovitis and bone edema were each scored from 0 (none/normal) to 3 (severe) at each joint. The total score for synovitis ranges from 0 to 36 and the total score for BME ranges from 0 to 72 since it is scored at both proximal and distal regions of each joint.
  The PsAMRIS composite score of BME and synovitis is calculated as: BME score + 2 × synovitis score. The score ranges from 0 (normal) to 144 (severe). Population: Full analysis set participants with available data.
  score on a scale
    number analyzed (Participants) | 114
    (all) | 15.12 (13.501)
Periarticular Inflammation Score Assessed by PsAMRIS [Mean (Standard Deviation); unit: score on a scale] — The OMERACT PsAMRIS scoring system assesses MCP, PIP, and DIP joints of fingers 2 to 5 of the most affected hand.
  Periarticular inflammation was scored 0 (absent) or 1 (present) separately at volar and dorsal aspects of the same 12 joint regions as evaluated for synovitis and flexor tenosynovitis. The score for periarticular inflammation ranges from 0 (absent) to 24 (present at all joints). Population: Full analysis set participants with available data.
  score on a scale
    number analyzed (Participants) | 115
    (all) | 2.47 (2.709)
Total Inflammation Score Assessed by PsAMRIS [Mean (Standard Deviation); unit: score on a scale] — The OMERACT PsAMRIS scoring system assesses MCP, PIP, and DIP joints of fingers 2 to 5 of the most affected hand. The PsAMRIS total inflammation score consists of BME, synovitis, tenosynovitis and periarticular inflammation.
  The total inflammation score is calculated as BME score + 2 × synovitis score + 2 × tenosynovitis + 3 × periarticular inflammation. The total inflammation score ranges from 0 (normal) to 288 (severe). Population: Full analysis set participants with available data.
  score on a scale
    number analyzed (Participants) | 114
    (all) | 25.79 (24.191)
Bone Erosion Score Assessed by PsAMRIS [Mean (Standard Deviation); unit: score on a scale] — The OMERACT PsAMRIS scoring system assesses bone erosion at the proximal and distal regions of MCP, PIP, and DIP joints of fingers 2 to 5 of the most affected hand.
  Bone erosion (loss of bone) was assessed on a scale of 0-10, based on the proportion of eroded bone compared to the assessed bone volume (articular surface to a depth of 1 cm), judged on all available images, where 0: no erosion; 1: 1-10% of bone eroded; 2: 11-20%, etc. The total bone erosion score is from 0 (none) to 240 (severe). Population: Full analysis set participants with available data.
  score on a scale
    number analyzed (Participants) | 115
    (all) | 2.19 (4.561)
Bone Proliferation Score Assessed by PsAMRIS [Mean (Standard Deviation); unit: score on a scale] — The OMERACT PsAMRIS scoring system assesses MCP, PIP, and DIP joints of fingers 2 to 5 of the most affected hand. Bone proliferation is abnormal bone formation in the periarticular region, such as at the entheses (enthesophytes) and across the joint (ankylosis).
  Bone proliferation was scored at each joint as 0 (absent) or 1 (present). The total bone proliferation score is from 0 (none) to 12 (present at all joints). Population: Full analysis set participants with available data.
  score on a scale
    number analyzed (Participants) | 115
    (all) | 2.32 (1.608)
Total Damage Score Assessed by PsAMRIS [Mean (Standard Deviation); unit: score on a scale] — The OMERACT PsAMRIS assesses MCP, PIP, and DIP joints of fingers 2 to 5 of the most affected hand. Erosion was assessed at distal and proximal regions of each joint from 0 to 10 based on the proportion of eroded bone compared to assessed bone volume. The total erosion score is from 0 to 240 (severe).
  Bone proliferation was scored at each joint as 0 (absent) or 1 (present); the total score is from 0 to 12 (worst).
  The total damage score consists of the erosion score and the bone proliferation score, calculated as: Erosion score + 20 × Bone Proliferation score, and ranges from 0 to 480 (worst). Population: Full analysis set participants with available data.
  score on a scale
    number analyzed (Participants) | 115
    (all) | 48.51 (35.147)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Composite Score of BME, Synovitis, and Tenosynovitis Assessed by PsAMRIS at Week 24
Description: PsAMRIS is a validated MRI scoring system that assesses metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints of fingers 2 to 5 of the most affected hand (the hand with the greater inflammatory burden of swollen joints and/or dactylitis).
  Synovitis, flexor tenosynovitis, and bone marrow edema were scored from 0 (none/normal) to 3 (severe) at each joint. The total scores for synovitis and tenosynovitis range from 0 to 36 and the total score for BME ranges from 0 to 72 since both proximal and distal regions of each joint were scored.
  The PsAMRIS composite inflammation score is calculated as: BME score + 2 × synovitis score + 2 × tenosynovitis score, and ranges from 0 (normal) to 216 (severe). A negative change from baseline indicates improvement.
  This endpoint was analyzed using a mixed-effects model for repeated measures (MMRM) with change from baseline as the dependent variable; baseline value, scanner type and time as independent variables.
Time Frame: Baseline and week 24
Population: Full analysis set participants with available data at baseline and week 24
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 98
score on a scale | -2.32 [-4.73 to 0.09]

2. Secondary Outcome: Change From Baseline in the Composite Score of BME, Synovitis, and Tenosynovitis Assessed by PsAMRIS at Week 48
Description: PsAMRIS is a validated MRI scoring system that assesses metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints of fingers 2 to 5 of the most affected hand (the hand with the greater inflammatory burden of swollen joints and/or dactylitis).
  Synovitis, flexor tenosynovitis, and bone marrow edema were scored from 0 (none/normal) to 3 (severe) at each joint. The total scores for synovitis and tenosynovitis range from 0 to 36 and the total score for BME ranges from 0 to 72 since both proximal and distal regions of each joint were scored.
  The PsAMRIS composite inflammation score is calculated as: BME score + 2 × synovitis score + 2 × tenosynovitis score, and ranges from 0 (normal) to 216 (severe). A negative change from baseline indicates improvement.
  This endpoint was analyzed using a MMRM with change from baseline as the dependent variable; baseline value, scanner type and time as independent variables.
Time Frame: Baseline and week 48
Population: Full analysis set participants with available data at baseline and week 48
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 81
score on a scale | -2.91 [-5.45 to -0.37]

3. Secondary Outcome: Change From Baseline in the Composite Score of BME and Synovitis Assessed by PsAMRIS at Weeks 24 and 48
Description: PsAMRIS is a validated MRI scoring system that assesses metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints of fingers 2 to 5 of the most affected hand (the hand with the greater inflammatory burden of swollen joints and/or dactylitis).
  Synovitis and bone marrow edema were each scored from 0 (none/normal) to 3 (severe) at each joint. The total score for synovitis ranges from 0 to 36 and the total score for BME ranges from 0 to 72 since this is scored at both proximal and distal regions of each joint.
  The PsAMRIS composite score of BME and synovitis is calculated as: BME score + 2 × synovitis score. The score ranges from 0 (normal) to 144 (severe). A negative change from baseline indicates improvement.
  This endpoint was analyzed using a MMRM including change from baseline of composite score of BME and synovitis as dependent variable; baseline value, scanner type and time as independent variables.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 98
score on a scale
  Week 24 | -1.19 [-2.89 to 0.50]
  Week 48: number analyzed (Participants) | 81
  Week 48 | -1.54 [-3.53 to 0.46]

4. Secondary Outcome: Change From Baseline in the PsAMRIS Total Inflammation Score at Weeks 24 and 48
Description: PsAMRIS is a validated MRI scoring system that assesses metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints of fingers 2 to 5 of the most affected hand.
  Synovitis, flexor tenosynovitis, and bone marrow edema were each scored from 0 (none/normal) to 3 (severe) at each joint. Periarticular inflammation was scored 0 (absent) or 1 (present) separately at volar and dorsal aspects of the same 12 joints. The scores for synovitis and tenosynovitis range from 0 to 36, the score for BME is from 0 to 72 and the periarticular inflammation score is from 0 to 24.
  The PsAMRIS total inflammation score is calculated as: BME score + 2 × synovitis score + 2 × tenosynovitis score + 3 × periarticular inflammation, and ranges from 0 (normal) to 288 (severe). A negative change from baseline indicates improvement.
  This endpoint was analyzed using a MMRM with change from baseline score as dependent variable; baseline value, scanner type and time as independent variables.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 98
score on a scale
  Week 24 | -3.62 [-7.11 to -0.12]
  Week 48: number analyzed (Participants) | 81
  Week 48 | -4.35 [-8.14 to -0.56]

5. Secondary Outcome: Change From Baseline in Bone Marrow Edema Assessed by PsAMRIS at Weeks 24 and 48
Description: Bone marrow edema (BME) is a buildup of fluid inside the bones. The OMERACT PsAMRIS scoring system assesses BME at the proximal and distal regions of MCP, PIP, and DIP joints of fingers 2 to 5 of the most affected hand. BME is assessed on a scale of 0-3 based on the proportion of bone with edema, compared to the assessed bone volume (articular surface to a depth of 1 cm), judged on all available images; where 0: no edema; 1: 1-33% of bone edema; 2: 34-66% of bone edema; 3: 67-100% of bone edema. The overall score ranges from 0 (none) to 72 (severe). A negative change from baseline indicates improvement.
  This endpoint was analyzed using a MMRM with change from baseline BME score as dependent variable; baseline value, scanner type and time as independent variables.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at weeks 24 and 48
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 99
score on a scale
  Week 24 | -0.22 [-0.83 to 0.38]
  Week 48: number analyzed (Participants) | 82
  Week 48 | -0.39 [-1.14 to 0.37]

6. Secondary Outcome: Change From Baseline in Synovitis Assessed by PsAMRIS at Weeks 24 and 48
Description: PsAMRIS is a validated MRI scoring system that assesses metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints of fingers 2 to 5 of the most affected hand (the hand with the greater inflammatory burden of swollen joints and/or dactylitis).
  Synovitis is inflammation of the synovial membrane, connective tissue that lines the inside of the joint.
  Synovitis was scored from 0 to 3 at MCP, PIP and DIP joints of fingers 2 to 5 (total of 12 joints), where score 0 is normal, and a score of 1 is mild, 2 is moderate, and 3 is severe. The overall synovitis score ranges from 0 (normal) to 36 (severe). A negative change from baseline indicates improvement.
  This endpoint was analyzed using a MMRM including change from baseline in synovitis score as dependent variable; baseline value, scanner type and time as independent variables.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 99
score on a scale
  Week 24 | -0.47 [-1.11 to 0.16]
  Week 48: number analyzed (Participants) | 82
  Week 48 | -0.65 [-1.39 to 0.10]

7. Secondary Outcome: Change From Baseline in Tenosynovitis Assessed by PsAMRIS at Weeks 24 and 48
Description: PsAMRIS is a validated MRI scoring system that assesses metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints of fingers 2 to 5 of the most affected hand (the hand with the greater inflammatory burden of swollen joints and/or dactylitis).
  Tenosynovitis is inflammation of the protective sheath (synovial membrane) that surrounds tendons.
  Flexor tenosynovitis was scored from 0 to 3 at MCP, PIP and DIP joints of fingers 2 to 5 (total of 12 joints) where a score of 0 is none; 1: < 1/2 tendon thickness; 2: ≥ 1/2 and < 1 tendon thickness; 3: ≥ 1 tendon thickness. The overall tenosynovitis score ranges from 0 (none) to 36 (severe). A negative change from baseline indicates improvement.
  This endpoint was analyzed using a MMRM including change from baseline in tenosynovitis score as dependent variable; baseline value, scanner type and time as independent variables.
Time Frame: Baseline and Weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 99
score on a scale
  Week 24 | -0.64 [-1.10 to -0.19]
  Week 48: number analyzed (Participants) | 82
  Week 48 | -0.78 [-1.15 to -0.40]

8. Secondary Outcome: Change From Baseline in Periarticular Inflammation Assessed by PsAMRIS at Weeks 24 and 48
Description: PsAMRIS is a validated MRI scoring system that assesses metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints of fingers 2 to 5 of the most affected hand (the hand with the greater inflammatory burden of swollen joints and/or dactylitis).
  Periarticular inflammation refers to inflammation of the tissues surrounding the joint, including the periosteum and the entheses, but not the tendon sheaths.
  Periarticular inflammation was scored 0 (absent) or 1 (present) separately at volar and dorsal aspects of the same 12 joint regions as evaluated for synovitis and flexor tenosynovitis. The score for periarticular inflammation ranges from 0 (absent) to 24 (present at all joints). A negative change from baseline indicates improvement.
  This endpoint was analyzed using a MMRM including change from baseline in periarticular inflammation as dependent variable; baseline value, scanner type and time as independent variables.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 99
score on a scale
  Week 24 | -0.49 [-0.90 to -0.07]
  Week 48: number analyzed (Participants) | 81
  Week 48 | -0.59 [-1.04 to -0.13]

9. Secondary Outcome: Change From Baseline in the PsAMRIS Total Damage Score at Weeks 24 and 48
Description: PsAMRIS is a validated MRI scoring system that assesses MCP, PIP, and DIP joints of fingers 2 to 5 of the most affected hand.
  Bone erosion (loss of bone) was assessed at the distal and proximal regions of each joint on a scale of 0 to 10, based on the proportion of eroded bone compared to the assessed bone volume, where 0 is no erosion; 1: 1-10% of bone eroded; 2: 11-20%, etc. The total erosion score is from 0 (none) to 240 (severe).
  Bone proliferation (abnormal bone formation in the periarticular region) was scored at each joint as 0 (absent) or 1 (present). The total proliferation score is from 0 to 12 (present at all joints) The total damage score includes the erosion and bone proliferation scores, calculated as: Erosion score + 20 × bone proliferation score, and ranges from 0 (none) to 480 (worst). A negative change from baseline indicates improvement.
  This endpoint was analyzed using a MMRM with baseline value, scanner type and time as independent variables.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 100
score on a scale
  Week 24 | 0.22 [-1.10 to 0.53]
  Week 48: number analyzed (Participants) | 83
  Week 48 | 0.50 [-0.38 to 1.38]

10. Secondary Outcome: Change From Baseline in Bone Erosion Assessed by PsAMRIS at Weeks 24 and 48
Description: PsAMRIS is a validated MRI scoring system that assesses metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints of fingers 2 to 5 of the most affected hand.
  Bone erosion (loss of bone) was assessed at the distal and proximal regions of each joint on a scale of 0-10, based on the proportion of eroded bone compared to the assessed bone volume, judged on all available images: 0: no erosion; 1: 1-10% of bone eroded; 2: 11-20%, etc. The assessed bone volume is from the articular surface (or its best estimated position if absent) to a depth of 1 cm. The total erosion score ranges from 0 (none) to 240 (severe). A negative change from baseline indicates improvement.
  This endpoint was analyzed using a MMRM with baseline value, scanner type and time as independent variables.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 100
score on a scale
  Week 24 | -0.01 [-0.06 to 0.05]
  Week 48: number analyzed (Participants) | 83
  Week 48 | 0.03 [-0.04 to 0.10]

11. Secondary Outcome: Change From Baseline in Bone Proliferation Assessed by PsAMRIS at Weeks 24 and 48
Description: PsAMRIS is a validated MRI scoring system that assesses metacarpophalangeal, proximal interphalangeal, and distal interphalangeal joints of fingers 2 to 5 of the most affected hand.
  Bone proliferation (abnormal bone formation in the periarticular region such as at the entheses and across the joint) was scored at each joint as 0 (absent) or 1 (present). The total proliferation score ranges from 0 (none) to 12 (present at all joints). A negative change from baseline indicates improvement.
  This endpoint was analyzed using a MMRM with baseline value, scanner type and time as independent variables.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 100
score on a scale
  Week 24 | 0.01 [-0.01 to 0.03]
  Week 48: number analyzed (Participants) | 83
  Week 48 | 0.02 [-0.02 to 0.07]

12. Secondary Outcome: Change From Baseline in Swollen Joint Count (SJC) at Weeks 24 and 48
Description: A total of 76 joints (including the distal interphalangeal joints of the fingers and toes) were examined for swelling.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Apremilast
Number analyzed (Participants) | 98
joints
  Week 24 | -5.8 (7.11)
  Week 48: number analyzed (Participants) | 81
  Week 48 | -6.3 (8.02)

13. Secondary Outcome: Change From Baseline in Tender Joint Count (TJC) at Weeks 24 and 48
Description: A total of 78 joints (including the distal interphalangeal joints of the fingers and toes) were examined for pain or tenderness.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Apremilast
Number analyzed (Participants) | 98
joints
  Week 24 | -7.9 (9.39)
  Week 48: number analyzed (Participants) | 81
  Week 48 | -8.4 (10.97)

14. Secondary Outcome: Change From Baseline in the Clinical Disease Activity Index for Psoriatic Arthritis (c-DAPSA) Score at Weeks 24 and 48
Description: The c-DAPSA is a measure of PsA disease activity, associated with functional and structural outcomes.
  C-DAPSA is calculated as the sum of the following measures:
  * Tender joint count 68 (TJC68);
  * Swollen joint count 66 (SJC66);
  * Patient global assessment of disease activity measured on a numerical rating scale (NRS) from 0 (not active) to 10 (very active); and
  * Pain measured on a NRS from 0 (none) to 10 (worst pain imaginable).
  The c-DAPSA score ranges from 0 to 154, where a higher score indicates greater disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 98
score on a scale
  Week 24 | -15.3 (14.04)
  Week 48: number analyzed (Participants) | 81
  Week 48 | -17.2 (16.46)

15. Secondary Outcome: Change From Baseline in Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index at Weeks 24 and 48 in Participants With Pre-existing Enthesopathy
Description: Enthesitis is inflammation of the sites where tendons or ligaments insert into the bone. The SPARCC Enthesitis Index assesses 16 unique sites for tenderness recorded as either present (1) or absent (0) for an overall score range of 0 to 16. A higher count represents greater enthesitis burden. A negative change from baseline indicates improvement.
  Pre-existing enthesopathy was defined as a baseline SPARCC score greater than 0.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with pre-existing enthesopathy (baseline SPARCC > 0) and available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 96
score on a scale
  Week 24 | -1.8 (2.26)
  Week 48: number analyzed (Participants) | 79
  Week 48 | -2.3 (2.00)

16. Secondary Outcome: Change From Baseline in the Leeds Enthesitis Index (LEI) at Weeks 24 and 48 in Participants With Pre-existing Enthesopathy
Description: LEI is a validated tool for the assessment of enthesitis in PsA patients. Tenderness was assessed at 6 sites of tendon insertion (lateral epicondyle, left and right, medial femoral condyle, left and right, and Achilles tendon insertion, left and right). Tenderness was recorded as either present (1) or absent (0) for each of the 6 sites, for an overall score range of 0 to 6. A higher count represents a greater enthesitis burden. A negative change from baseline indicates improvement.
  Pre-existing enthesopathy was defined as a baseline LEI score greater than 0.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with pre-existing enthesopathy (baseline LEI > 0) and available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 78
score on a scale
  Week 24 | -1.3 (1.38)
  Week 48: number analyzed (Participants) | 61
  Week 48 | -1.5 (1.19)

17. Secondary Outcome: Percentage of Participants With Baseline SPARCC Enthesitis Whose Enthesitis Improved to 0 at Weeks 24 and 48
Description: Enthesitis is inflammation of the sites where tendons or ligaments insert into the bone. The SPARCC Enthesitis Index assesses 16 unique sites for tenderness recorded as either present (1) or absent (0) for an overall score range of 0 to 16. A higher count represents greater enthesitis burden. Resolution of SPARCC enthesitis is defined as achieving a SPARCC index score of 0 for participants with baseline SPARCC enthesitis (SPARCC index score > 0).
Time Frame: Weeks 24 and 48
Population: Full analysis set participants with SPARCC enthesitis at baseline (SPARCC score > 0) and non-missing SPARCC scores at each time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast
Number analyzed (Participants) | 96
percentage of participants
  Week 24 | 46.9 [36.61 to 57.34]
  Week 48: number analyzed (Participants) | 79
  Week 48 | 57.0 [45.33 to 68.06]

18. Secondary Outcome: Percentage of Participants With Baseline LEI Enthesitis Whose Enthesitis Improved to 0 at Weeks 24 and 48
Description: LEI is a validated tool for the assessment of enthesitis in PsA patients. Tenderness was assessed at 6 sites of tendon insertion (lateral epicondyle, left and right, medial femoral condyle, left and right, and Achilles tendon insertion, left and right). Tenderness was recorded as either present (1) or absent (0) for each of the 6 sites, for an overall score range of 0 to 6. A higher count represents a greater enthesitis burden. Resolution of LEI enthesitis is defined as a LEI score of 0 for participants with baseline LEI enthesitis (LEI score > 0).
Time Frame: Weeks 24 and 48
Population: Full analysis set participants with LEI enthesitis at baseline (LEI score > 0) and non-missing LEI scores at each time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast
Number analyzed (Participants) | 78
percentage of participants
  Week 24 | 56.4 [44.70 to 67.61]
  Week 48: number analyzed (Participants) | 61
  Week 48 | 62.3 [48.96 to 74.39]

19. Secondary Outcome: Change From Baseline in Leeds Dactylitis Index (LDI) at Weeks 24 and 48 in Participants With Pre-existing Dactylitis
Description: Dactylitis is characterized by the swelling of the entire finger or toe. Dactylitis was assessed using the Leeds Dactylitis Index (LDI). LDI measures the ratio of the circumference of the affected digit to the circumference of the digit on the opposite hand or foot, using a minimum difference of 10% to define a dactylitic digit. The ratio of circumference is multiplied by a tenderness score from 0 to 3, where 0 = No Tenderness, 1 = Tender, 2 = Tender and wince, 3 = Tender and withdraw. The dactylitis score is the sum of the individual scores for each digit, where 0 indicates no dactylitis and higher scores represent worse dactylitis. A negative change from baseline indicates improvement.
  Pre-existing dactylitis is defined as a baseline LDI score greater than 0.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with pre-existing dactylitis (LDI > 0) and available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 37
score on a scale
  Week 24 | -34.38 (21.322)
  Week 48: number analyzed (Participants) | 30
  Week 48 | -38.71 (21.793)

20. Secondary Outcome: Percentage of Participants With Baseline Dactylitis Whose Dactylitis Count Improved to 0 at Weeks 24 and 48
Description: Dactylitis is characterized by the swelling of the entire finger or toe. Dactylitis was assessed using the Leeds Dactylitis Index (LDI). LDI measures the ratio of the circumference of the affected digit to the circumference of the digit on the opposite hand or foot, using a minimum difference of 10% to define a dactylitic digit. The ratio of circumference is multiplied by a tenderness score from 0 to 3 , where 0 = No Tenderness, 1 = Tender, 2 = Tender and wince, 3 = Tender and withdraw). The LDI score is the sum of the individual scores for each digit, where 0 is no dactylitis and higher scores represent worse dactylitis.
  Resolution of dactylitis is defined as a LDI score of 0 for participants with dactylitis (LDI score > 0) at baseline.
Time Frame: Weeks 24 and 48
Population: Full analysis set participants with dactylitis at baseline (LDI > 0) and non-missing LDI scores at each time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apremilast
Number analyzed (Participants) | 37
percentage of participants
  Week 24 | 89.2 [74.58 to 96.97]
  Week 48: number analyzed (Participants) | 30
  Week 48 | 93.3 [77.93 to 99.18]

21. Secondary Outcome: Change From Baseline in the Psoriatic Arthritis Disease Activity Score (PASDAS) at Weeks 24 and 48
Description: PASDAS is a measure of disease activity derived from the following variables:
  * Physician and patient global assessment of disease activity (assessed on a 0-10 NRS, then multiplied by 10)
  * 68 tender joint count
  * 66 swollen joint count
  * Short Form-36 Questionnaire (SF-36) physical component summary score (general health status on a scale from 0-100)
  * Tender dactylitis count (each digit assessed for tender dactylitis; total score 0-20)
  * Leeds enthesitis index (enthesitis assessed at 6 sites; total score of 0-6)
  * C-reactive protein (CRP) level (mg/L) The composite score is a weighted index that ranges from 0 to 10, with worse disease activity represented by higher scores. A negative change from baseline indicates improvement.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 103
score on a scale
  Week 24 | -1.752 (1.3002)
  Week 48: number analyzed (Participants) | 88
  Week 48 | -1.833 (1.4146)

22. Secondary Outcome: Change From Baseline in the Evaluator's Global Assessment of Disease Activity at Weeks 24 and 48
Description: The Evaluator's Global Assessment of Disease Activity evaluates how active a participant's PsA was on the day of the assessment. Disease activity was assessed on a 0 to 10 numeric rating scale (NRS) where 0 represents "no arthritis activity," and 10 represents "extreme active arthritis". A negative change from baseline indicates improvement.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 98
score on a scale
  Week 24 | -2.7 (1.99)
  Week 48: number analyzed (Participants) | 81
  Week 48 | -2.8 (2.11)

23. Secondary Outcome: Change From Baseline in the Patient's Global Assessment of Disease Activity at Weeks 24 and 48
Description: The Patient's Global Assessment is an assessment of how active a participant's arthritis was on average during the past week. The score ranges from 0 to 10 based on a numerical rating scale, where 0 represents 'Very Well' and 10 represents 'Very Poor'. A negative change from baseline indicates improvement.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 99
score on a scale
  Week 24 | -1.3 (2.09)
  Week 48: number analyzed (Participants) | 82
  Week 48 | -1.6 (2.24)

24. Secondary Outcome: Change From Baseline in the Subject's Assessment of Pain at Weeks 24 and 48
Description: The Subject's Assessment of Pain is an assessment of how much pain a participant had on average during the past week due to psoriatic arthritis. The score ranges from 0-10 based on a numerical rating scale, where 0 represents 'No Pain' and 10 represents 'Pain As Bad As You Can Imagine'. A negative change from baseline indicates improvement.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 99
score on a scale
  Week 24 | -1.4 (2.10)
  Week 48: number analyzed (Participants) | 82
  Week 48 | -2.0 (2.13)

25. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) at Weeks 24 and 48
Description: The Health Assessment Questionnaire Disability Index is a patient-reported questionnaire that measures the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores) over the past week. Participants assessed their ability to do each task on a scale from 0 (without any difficulty) to 3 (unable to do). Scores were averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 represents very severe, high-dependency disability. A negative change from Baseline in the overall score indicates improvement.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 99
score on a scale
  Week 24 | -0.293 (0.4162)
  Week 48: number analyzed (Participants) | 82
  Week 48 | -0.383 (0.4654)

26. Secondary Outcome: Change From Baseline in Whole Body MRI (WB-MRI) Peripheral Enthesitis Inflammation Index at Weeks 24 and 48
Description: Enthesitis was assessed by whole body MRI according to the OMERACT MRI Whole-Body Score for Inflammation in Peripheral Joints and Entheses in Inflammatory Arthritis (MRI-WIPE) scoring system. Thirty-three entheseal sites were assessed for soft tissue inflammation (STI) and 34 sites for osteitis, including the shoulder, pelvis, knees and feet, each on a scale from 0 (none) to 3 (severe).
  The Total Peripheral Enthesitis Inflammation score is calculated by adding up all the enthesitis (STI and osteitis) scores and ranges from 0 to 201, with higher scores reflecting greater disease severity. A negative change from baseline indicates improvement.
  WB-MRI endpoints were analyzed using a MMRM including change from baseline as dependent variable; baseline value, scanner type and time as independent variables.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 100
score on a scale
  Week 24 | -0.17 [-0.65 to 0.31]
  Week 48: number analyzed (Participants) | 84
  Week 48 | -0.52 [-1.01 to -0.02]

27. Secondary Outcome: Change From Baseline in the WB-MRI Peripheral Joints Inflammation Index at Weeks 24 and 48
Description: Joint inflammation was assessed by whole body MRI according to the OMERACT MRI-WIPE scoring system. Eighty-three peripheral joints were assessed for synovitis and 96 sites for osteitis at the shoulder, hands, pelvis, knees and feet on a semiquantitative scale from 0 (none) to 3 (severe).
  The Peripheral Joint Inflammation score is calculated by adding up all the joint (synovitis and osteitis) scores and ranges from 0 to 537, with higher scores reflecting greater disease severity. A negative change from baseline indicates improvement.
  WB MRI endpoints were analyzed using a MMRM including change from baseline as dependent variable; baseline value, scanner type and time as independent variables.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 100
score on a scale
  Week 24 | -3.38 [-5.10 to -1.66]
  Week 48: number analyzed (Participants) | 84
  Week 48 | -3.58 [-5.66 to -1.51]

28. Secondary Outcome: Change From Baseline in the WB-MRI Total Peripheral Inflammation Index at Weeks 24 and 48
Description: Inflammation in joints (arthritis) and at entheses (enthesitis) were assessed separately for soft tissues (synovitis at joints, soft tissue inflammation at entheses) and bone (osteitis) by whole body MRI according to the OMERACT MRI-WIPE scoring system. Each entheseal and joint was scored on a scale from 0 (none) to 3 (severe).
  The total peripheral inflammation index is the sum of peripheral enthesitis and peripheral joints inflammation index scores, and ranges from 0 to 738, with higher scores reflecting greater disease severity. A negative change from baseline indicates improvement.
  WB MRI endpoints were analyzed using a MMRM including change from baseline as dependent variable; baseline value, scanner type and time as independent variables.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 100
score on a scale
  Week 24 | -3.49 [-5.46 to -1.52]
  Week 48: number analyzed (Participants) | 84
  Week 48 | -4.06 [-6.39 to -1.72]

29. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Weeks 24 and 48
Description: BASDAI is a composite score based on a self-administered survey of six questions with each answered on a 0 to 10 NRS. The 6 questions assess the five major symptoms relevant to spondyloarthropathies: 1) fatigue; 2) spinal pain; 3) peripheral joint pain/swelling; 4) areas of localized tenderness; 5a) morning stiffness severity upon wakening; 5b) morning stiffness duration upon wakening.
  To give each of the 5 symptoms equal weighting, the mean of the two scores relating to morning stiffness (questions 5 and 6) is taken. The final BASDAI score is calculated as the mean of the 5 items. The BASDAI score ranges from 0 to 10, with higher scores reflecting greater disease activity. A negative change from baseline indicates improvement.
  BASDAI was analyzed in participants deemed to have PsA spondylitis by the investigator and with BASDAI item 2 score ≥ 4 at baseline).
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants deemed to have PsA spondylitis by the investigator and with BASDAI item 2 score ≥ 4 at baseline, and with available data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 35
score on a scale
  Week 24 | -1.94 (1.935)
  Week 48: number analyzed (Participants) | 31
  Week 48 | -2.01 (2.246)

30. Secondary Outcome: Change From Baseline in the Psoriatic Arthritis Impact of Disease 12 Domain Questionnaire (PsAID-12) at Weeks 24 and 48
Description: The PsAID consists of 12 physical and psychological domains: pain, fatigue, skin, work and/or leisure activities, function, discomfort, sleep, coping, anxiety, embarrassment and/or shame, social life, and depression.
  Each domain is scored on a NRS rom 0 to 10. The final score is derived as a weighted sum of each domain score, divided by 20, and has a range from 0 (best status) to 10 (worst status). A negative change from baseline indicates improvement.
Time Frame: Baseline and weeks 24 and 48
Population: Full analysis set participants with available data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast
Number analyzed (Participants) | 104
score on a scale
  Week 24 | -1.352 (1.8441)
  Week 48: number analyzed (Participants) | 90
  Week 48 | -1.612 (1.6613)

31. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE is any adverse event (AE) that began or worsened on or after the first dose of apremilast and no later than 28 days after the last dose.
  A serious adverse event is any AE occurring at any dose that:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly/birth defect;
  * Constituted an important medical event.
  For each AE, the Investigator assessed the severity/intensity of the event as mild, moderate, or severe (symptoms causing severe discomfort/pain, interference with daily activities, and requiring medical, surgical or drug therapy). The Investigator also assessed whether each event was suspected to be related to study drug based on whether there was evidence to suggest a causal relationship.
Time Frame: From first dose of study drug up to 28 days after last dose; up to 52 weeks.
Population: All participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast
Number analyzed (Participants) | 122
Participants
  Any treatment-emergent adverse event (TEAE) | 95
  Any drug-related TEAE | 60
  Any severe TEAE | 6
  Any serious TEAE | 6
  Any serious drug-related TEAE | 0
  Any TEAE leading to study drug interruption | 12
  Any TEAE leading to study drug withdrawal | 15
  Any TEAE leading to death | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 days after last dose; up to 52 weeks.
Description: All-cause mortality is reported for all enrolled participants. Adverse events are reported for all participants who received at least one dose of study drug.
Arm/Group | Apremilast
All-Cause Mortality (participants affected / at risk) | 0/123
Serious Adverse Events (participants affected / at risk) | 6/122
Other Adverse Events (participants affected / at risk) | 63/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apremilast (N=122)
Angina pectoris (Cardiac disorders) | 1
Non-cardiac chest pain (General disorders) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apremilast (N=122)
Diarrhoea (Gastrointestinal disorders) | 41
Dyspepsia (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 15
Nasopharyngitis (Infections and infestations) | 9
Headache (Nervous system disorders) | 13
Psoriasis (Skin and subcutaneous tissue disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT03783026/Prot_002.pdf
  • Statistical Analysis Plan (2022-05-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT03783026/SAP_003.pdf